CLINICAL TRIAL: NCT03152513
Title: A Combined Retrospective and Prospective Review of "Anesthesia Stat!" Events in the Pediatric Operating Room
Brief Title: A Review of "Anesthesia Stat!" in the Pediatric Operating Room
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00042123
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; Surgery; Critical Illness; Critical Incident
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to look at critical events in the pediatric operating room in a retrospective and now prospective fashion to determine if there are any trends such as age, presence of URI, type of surgery, type of airway, level of hands on provider, or other predictive markers associated these events so that we may gain some insight into perhaps reducing the incidence of these events or simply be more attune to the increased risks in certain situations.

DETAILED DESCRIPTION:
The goal of this study is to further characterize these events, determine the incidence in the operating room, unmask associated issues to improve vigilance, and to look and see if there are possibly improvements to be made in the investigators care of all pediatric patients to further reduce the incidence or sequelae of these events.

Also, the investigators want to characterize the details associated with these events. Do these patients have prolonged PACU stays? How long are these events? Are they mostly respiratory in nature? What is the average level of desaturation when it occurs. Is it primarily at the beginning, middle, or end of procedures.

This study will have a two pronged approach as the investigators have been collecting prospective observational data already for the QI project looking at this issue using the data sheet in Appendix 1. The investigators have been collecting this data since April of 2015 to the present. This data needs to be entered into a data base so that it can be analyzed in greater detail.

In addition to reviewing the data we have already obtained we would like to begin to collect data prospectively to add to the data we have already collected. Patients that have already been collected will assigned a study number based on the chronology of their event will older event receiving a smaller study ID number and more recent patient receiving a higher study number. This same sequence will continue into our prospective data base.

Going forward, the investigators will continue the current methodology of having study personnel who are present in the pediatric operating room respond to stat calls within the pediatric OR or other pediatric anesthetizing site. The study personnel will assist the practioner or practioners already present first, and when possible will collect data related to the event in real time or immediately afterward and enter that on the study data form.

The investigators will record basic demographic data about the patient including age, weight, height, presence of URI or Asthma, procedure, surgeon. The investigators will record the time of the event, duration, significant changes in vital signs, practitioners opinion of causality if possible, and any therapeutic steps that were instituted such as the administration of other medications, assistance with breathing, administration of oxygen, reintubation. This will be documented in the narrative section of the data sheet.

These data sheets will then have most data entered on them into a deidentified spread sheet. A linkage file will be created so that a patient's study ID can be linked to their actual medical record number in case other information would be necessary or helpful in further evaluating the "Anesthesia Stat," event already noted.

Study personnel will also review the narratives of these cases to determine if there are any common patterns that may not be readily apparent with simple numerical and case data entered into the database.

ELIGIBILITY:
Inclusion Criteria:

* Patients <18 years of age
* Patients undergoing anesthesia and/or surgery or a diagnostic procedure in the operating room or other anesthetizing sites for which a stat page for help has been initiated.

Exclusion Criteria:

* Patients >=18 years of age.
* Patients having a critical event not under anesthesia in other venues within Brenner's Children's hospital or within the pediatric intensive care unit.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects under the age of 18 are included in the study only after an "Anesthesia Stat," or overhead call for help has been initiated by the provider in the room or other nursing or operating room staff involved in that patient's care. Data will only be taken when a member of the study staff is present which is typically during the week, during the typical OR day, and not the weekends or late at night.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
The incidence of "Anesthesia Stat" critical events | 7 years
  The number of new cases of "Anesthesia Stat" critical events per population at risk in the study period

SECONDARY OUTCOMES:
Age of patients on which "Anesthesia Stat" has been called | 7 years
  Median Age in months of patients on which "Anesthesia Stat" has been called.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Pediatric Operating Room, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No